CLINICAL TRIAL: NCT01134614
Title: A Phase II Trial of GM-CSF Protein Plus Ipilimumab in Patients With Advanced Melanoma
Brief Title: Ipilimumab With or Without Sargramostim in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02039; NCI-2011-02039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000671238; E1608; 11-01460; E1608 (Other: ECOG-ACRIN Cancer Research Group); E1608 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2010-04-27; First posted 2010-06-02 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Melanoma; Metastatic Melanoma; Recurrent Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (ipilimumab and sargramostim) (Experimental): Patients receive induction therapy comprising ipilimumab IV over 90 minutes on day 1 and sargramostim SC once daily on days 1-14. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, anti-tumor response is assessed and patients then receive maintenance therapy comprising ipilimumab IV over 90 minutes on day 1 and sargramostim SC once daily on days 1-14. Treatment with ipilimumab repeats every 12 weeks and treatment with sargramostim repeats every 21 days. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy until disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Sargramostim
- Arm B (ipilimumab) (Active Comparator): Patients receive induction therapy comprising ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, anti-tumor response is assessed and patients then receive maintenance therapy of ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 12 weeks. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
  Arms: Arm A (ipilimumab and sargramostim)

SUMMARY:
This randomized phase II trial is studying how well giving ipilimumab with or without sargramostim (GM-CSF) works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery (unresectable). Ipilimumab works by activating the patient's immune system to fight cancer. Colony-stimulating factors, such as sargramostim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of treatment. It is not yet known whether giving ipilimumab together with sargramostim is more effective than ipilimumab alone in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall survival for the combination of sargramostim (GM-CSF) plus ipilimumab and ipilimumab alone in patients with advanced melanoma.

SECONDARY OBJECTIVES:

I. To evaluate the progression-free survival, response rate, safety and tolerability for the combination of GM-CSF plus ipilimumab and ipilimumab alone in patients with advanced melanoma.

II. To explore the utility of immune related response criteria (irRC) prospectively in patients receiving ipilimumab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive induction therapy comprising ipilimumab intravenously (IV) over 90 minutes on day 1 and sargramostim subcutaneously (SC) once daily on days 1-14. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, anti-tumor response is assessed and patients then receive maintenance therapy comprising ipilimumab IV over 90 minutes on day 1 and sargramostim SC once daily on days 1-14. Treatment with ipilimumab repeats every 12 weeks and treatment with sargramostim repeats every 21 days. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy until disease progression or unacceptable toxicity.

ARM B: Patients receive induction therapy comprising ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, anti-tumor response is assessed and patients then receive maintenance therapy of ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 12 weeks. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All sites of disease must be evaluated within 4 weeks prior to randomization; patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* No more than one prior systemic therapeutic regimen for unresectable stage III or stage IV melanoma; this includes chemotherapy, biologic therapy, biochemotherapy, or investigational treatment; this does not include any therapies given in the adjuvant setting
* Histologic diagnosis of metastatic melanoma; for unknown primary disease, diagnosis of metastatic disease by cytology fine needle aspiration (FNA) is not acceptable
* Women must not be pregnant or breast-feeding due to unknown effects of ipilimumab and GM-CSF on the unborn fetus; all women of childbearing potential must have a blood test within 72 hours prior to randomization to rule out pregnancy; women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception; women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized; sexually mature females who have not undergone a hysterectomy or who have not been postmenopausal naturally for at least 24 consecutive months (i.e., who have had menses at some time in the preceding 24 consecutive months) are considered to be of childbearing potential; women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential
* White blood cells (WBC) >= 2000/uL (obtained =< 4 weeks prior to randomization)
* Absolute neutrophil count (ANC) >= 1500/mcL (obtained =< 4 weeks prior to randomization)
* Platelets >= 100,000/mcL (obtained =< 4 weeks prior to randomization)
* Hemoglobin >= 8 g/dL (obtained =< 4 weeks prior to randomization)
* Creatinine =< 3.0 x upper limit of normal (ULN) (obtained =< 4 weeks prior to randomization)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (obtained =< 4 weeks prior to randomization)
* Bilirubin =< 3.0 x ULN, (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL) (obtained =< 4 weeks prior to randomization)
* No concomitant therapy with any of the following: interleukin (IL) 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids; must have been discontinued >= 4 weeks
* No infection with human immunodeficiency virus (HIV); due to the mechanism of action of ipilimumab and GM-CSF, activity and side effects in an immune compromised patient are unknown
* No active infection with hepatitis B
* No active or chronic infection with hepatitis C
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Patients with any history of central nervous system (CNS) metastases are excluded
* Patients are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Patients are excluded if they have a history of any autoimmune disease; patients with a history of autoimmune thyroiditis are eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy
* Patients are excluded for any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea
* Patients are excluded for receiving any non-oncology vaccine therapy used for prevention of infectious diseases for up to four weeks (28 days) prior to or after any dose of ipilimumab
* Patients are excluded if they have a history of prior treatment with ipilimumab or prior cluster of differentiation (CD)137 agonist or cytotoxic T-lymphocyte antigen 4 (CTLA-4) inhibitor or agonist
* Any concurrent medical condition requiring the use of systemic steroids is not permitted (the use of inhaled or topical steroids is permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2010-12-28 (Actual); Primary Completion 2013-02-15 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Frank S Hodi, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (258):
- United States (258):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Rush-Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Trinity Medical Center, Moline, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - San Juan Oncology Associates, Farmington, New Mexico
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Hodi FS, Lee S, McDermott DF, Rao UN, Butterfield LH, Tarhini AA, Leming P, Puzanov I, Shin D, Kirkwood JM. Ipilimumab plus sargramostim vs ipilimumab alone for treatment of metastatic melanoma: a randomized clinical trial. JAMA. 2014 Nov 5;312(17):1744-53. doi: 10.1001/jama.2014.13943. PMID 25369488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from ECOG member institutions between December 28, 2010 and July 28, 2011.
Groups:
- Arm A (Ipilimumab and Sargramostim): ARM A: Patients receive induction therapy comprising ipilimumab intravenously (IV) over 90 minutes on day 1 and sargramostim subcutaneously (SC) once daily on days 1-14. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, anti-tumor response is assessed and patients then receive maintenance therapy comprising ipilimumab IV over 90 minutes on day 1 and sargramostim SC once daily on days 1-14. Treatment with ipilimumab repeats every 12 weeks and treatment with sargramostim repeats every 21 days. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy until disease progression or unacceptable toxicity.
  ipilimumab: Given IV
  sargramostim: Given SC
- Arm B (Ipilimumab): ARM B: Patients receive induction therapy comprising ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, anti-tumor response is assessed and patients then receive maintenance therapy of ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 12 weeks. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  ipilimumab: Given IV
Period: Overall Study
Arm/Group | Arm A (Ipilimumab and Sargramostim) | Arm B (Ipilimumab)
Started | 123 | 122
Treated | 119 | 121
Treated and Toxicity Assessed | 118 | 120
Completed | 0 (Treatment continues until disease progression or unacceptable toxicity.) | 0 (Treatment continues until disease progression or unacceptable toxicities)
Not Completed | 123 | 122
Not completed — Still on treatment as of March 2013 | 21 | 13
Not completed — Progressive disease | 60 | 54
Not completed — Adverse Event | 26 | 39
Not completed — Death | 5 | 8
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Alternative therapy | 2 | 0
Not completed — Complicating disease | 2 | 1
Not completed — Physician's decision | 0 | 1
Not completed — Never started treatment | 4 | 1
Not completed — Pt received tx not allowed on study | 0 | 1
Not completed — Symptomatic deterioration | 0 | 1
Not completed — Patient in hospice care | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in this analysis.
Groups:
- Arm A (Ipilimumab and Sargramostim): ARM A: Patients receive induction therapy comprising ipilimumab intravenously (IV) over 90 minutes on day 1 and sargramostim subcutaneously (SC) once daily on days 1-14. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, patients then receive maintenance therapy comprising ipilimumab IV over 90 minutes on day 1 and sargramostim SC once daily on days 1-14. Treatment with ipilimumab repeats every 12 weeks and treatment with sargramostim repeats every 21 days. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy until disease progression or unacceptable toxicity.
  ipilimumab: Given IV
  sargramostim: Given SC
- Arm B (Ipilimumab): ARM B: Patients receive induction therapy comprising ipilimumab as in arm A. Patients then receive maintenance therapy comprising ipilimumab IV as in arm A. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy comprising ipilimumab IV as in arm A. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  ipilimumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm A (Ipilimumab and Sargramostim) | Arm B (Ipilimumab) | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 86] | 64 [21 to 89] | 63 [21 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 44 | 82
  Male | 85 | 78 | 163
Region of Enrollment [Number; unit: participants]
  United States | 123 | 122 | 245

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death from any cause.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ipilimumab and Sargramostim) | Arm B (Ipilimumab)
Number analyzed (Participants) | 123 | 122
Months | 17.5 [14.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 12.7 [10.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from randomization to disease progression or death, whichever occurs first. Response and disease progression will be evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Disease progression is defined as >= 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) and the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions is also considered progression.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ipilimumab and Sargramostim) | Arm B (Ipilimumab)
Number analyzed (Participants) | 123 | 122
Months | 3.1 [2.9 to 4.6] | 3.1 [2.9 to 4.0]

3. Secondary Outcome: Proportion of Patients With Objective Response
Description: Objective response was evaluated using RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 criteria. Per RECIST criteria, complete response (CR) = disappearance of all target and non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Partial response (PR)= At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. To be assigned a status of partial response, changes in tumor measurements must be confirmed by a repeat assessment performed no less than four weeks after the criteria for response is met. Objective response = CR + PR.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years
Population: All randomized patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Ipilimumab and Sargramostim) | Arm B (Ipilimumab)
Number analyzed (Participants) | 123 | 122
Proportion of patients | 0.155 [0.096 to 0.231] | 0.148 [0.090 to 0.223]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Arm A (Ipilimumab and Sargramostim): ARM A: Patients receive induction therapy comprising ipilimumab intravenously (IV) over 90 minutes on day 1 and sargramostim subcutaneously (SC) once daily on days 1-14. Treatment repeats every 21 days for 4 cycles. After 12 weeks of induction treatment, patients then receive maintenance therapy comprising ipilimumab IV over 90 minutes on day 1 and sargramostim SC once daily on days 1-14. Treatment with ipilimumab repeats every 12 weeks and treatment with sargramostim repeats every 21 days. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy until disease progression or unacceptable toxicity.
- Arm B (Ipilimumab): ARM B: Patients receive induction therapy comprising ipilimumab as in arm A. Patients then receive maintenance therapy comprising ipilimumab IV as in arm A. After 12 weeks of maintenance therapy, anti-tumor response is reassessed and patients with responsive or stable disease then continue maintenance therapy comprising ipilimumab IV as in arm A. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Ipilimumab and Sargramostim) | Arm B (Ipilimumab)
Serious Adverse Events (participants affected / at risk) | 56/118 | 69/120
Other Adverse Events (participants affected / at risk) | 110/118 | 111/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipilimumab and Sargramostim) (N=118) | Arm B (Ipilimumab) (N=120)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 7 | 4
Fever (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 0 | 1
Injection site reaction (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 11
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Colitis (Gastrointestinal disorders) | 7 | 12
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 2 | 7
Diarrhea (Gastrointestinal disorders) | 14 | 15
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 0 | 5
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 1
Kidney infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Activated PTT prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 8
Alkaline phosphatase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 5 | 9
Blood bilirubin increased (Investigations) | 0 | 4
Creatinine increased (Investigations) | 1 | 0
INR increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 6 | 6
Lymphocyte count decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 2 | 2
Serum amylase increased (Investigations) | 2 | 1
White blood cell decreased (Investigations) | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipilimumab and Sargramostim) (N=118) | Arm B (Ipilimumab) (N=120)
Anemia (Blood and lymphatic system disorders) | 22 | 24
Chills (General disorders) | 18 | 8
Edema limbs (General disorders) | 10 | 4
Fatigue (General disorders) | 70 | 75
Fever (General disorders) | 17 | 18
Injection site reaction (General disorders) | 62 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 50 | 54
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 62 | 57
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 7 | 1
Adrenal insufficiency (Endocrine disorders) | 7 | 2
Hypothyroidism (Endocrine disorders) | 11 | 6
Abdominal pain (Gastrointestinal disorders) | 20 | 16
Constipation (Gastrointestinal disorders) | 7 | 9
Diarrhea (Gastrointestinal disorders) | 46 | 46
Nausea (Gastrointestinal disorders) | 36 | 31
Vomiting (Gastrointestinal disorders) | 10 | 6
Alanine aminotransferase increased (Investigations) | 13 | 18
Alkaline phosphatase increased (Investigations) | 12 | 12
Aspartate aminotransferase increased (Investigations) | 16 | 21
Blood bilirubin increased (Investigations) | 6 | 6
Creatinine increased (Investigations) | 6 | 8
Lipase increased (Investigations) | 13 | 7
Lymphocyte count decreased (Investigations) | 6 | 9
Platelet count decreased (Investigations) | 9 | 4
Weight loss (Investigations) | 16 | 17
Investigations - Other, specify (Investigations) | 7 | 7
Anorexia (Metabolism and nutrition disorders) | 25 | 33
Hyperuricemia (Metabolism and nutrition disorders) | 6 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 2
Hyponatremia (Metabolism and nutrition disorders) | 9 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1
Dizziness (Nervous system disorders) | 11 | 5
Dysgeusia (Nervous system disorders) | 7 | 7
Headache (Nervous system disorders) | 23 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Hot flashes (Vascular disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less